CLINICAL TRIAL: NCT02999802
Title: Nutrient Sensing & Signaling in Aging Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-0226; R56AG051267 (NIH)
Record Dates: First submitted 2016-12-09; First posted 2016-12-21 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2017-08

CONDITIONS: Nutrient Sensing
Keywords: Nutrient Sensing; Exercise; Elderly
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise (Experimental): Determining the effect of 12 weeks of resistance training exercise on the response of muscle amino acid sensing
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Progressive resistance exercise training

SUMMARY:
This research seeks to better understand how cellular and molecular bases of changes associated with aging contribute to decreased function and increased incidence of disease. Specific mechanism in muscle responsible for anabolic resistance - a key component of sarcopenia and frailty - will be identified. The proposed research is relevant to public health because the discovery of new targets for interventions and novel therapeutics to improve muscle strength and function, prevent falls, and reduce physical dependency will improve the healthspan and quality of life in older adults by improving their physical function and ability to remain independent and healthy for a longer period of time.

DETAILED DESCRIPTION:
Anabolic resistance to nutrition is the reduced ability of skeletal muscle to increase protein synthesis in response to feeding. It is a major contributor to muscle atrophy in aging, inactivity, burns, trauma, and cancer cachexia. The effects of anabolic resistance on health and physical function are important. For example, the loss of muscle mass and strength with aging (sarcopenia) increases the risk for falls, physical dependency and morbidity in older adults. A major determinant of muscle size is muscle protein content, which is controlled by the fine balance between protein synthesis and breakdown. Recently, investigators have found that amino acids and exercise independently increase muscle protein synthesis and overall anabolism by activating the mammalian/mechanistic target of rapamycin complex 1 (mTORC1) signaling pathway in humans. Aging and inactivity reduce these anabolic effects, but the underlying mechanisms of anabolic resistance are not known. The purpose of this application is to better understand how anabolic resistance develops in skeletal muscle. The long-term goal is to identify specific molecular targets for the development of evidence-based clinical interventions to counteract anabolic resistance and muscle wasting in clinical populations. Here, investigators will focus on one potential mechanisms underlying anabolic resistance to amino acids: activation of mTORC1 in human muscle cells. The central hypothesis is that the physical activity restores mTORC1 signaling which is the primary contributor to anabolic resistance in human skeletal muscle. Investigators will test this hypothesis in healthy subjects with the following specific aim: Determine the effect of increasing habitual physical activity on anabolic resistance. Investigators will study human subjects utilizing stable isotopes model to measure amino acid kinetics and muscle protein metabolism in combination with molecular analysis of muscle to determine the regulatory role of amino acids, physical inactivity, and amino acid transporter functional activity on mTORC1. The proposed approach is innovative because it represents a new and substantial departure from the status quo as investigators will examine the underlying mechanisms of anabolic resistance to nutrition using novel methodological approaches. The proposed research is significant because it will lead to the development of evidence-based interventions to treat sarcopenia and muscle wasting.

ELIGIBILITY:
Inclusion Criteria:

* 65-80 yrs
* Stable body weight for at least 1 year
* Ability to sign consent form:

Exclusion Criteria:

* Exercise training (>2 weekly sessions of moderate to high intensity aerobic or resistance exercise)
* Physical dependence or frailty (impairment in the Activities of Daily Living (ADL), history of falls (>2/year), or >5% weight loss in the past year)
* Significant heart, liver, kidney, blood, or respiratory disease
* Peripheral vascular disease
* Diabetes mellitus or other untreated endocrine disease
* Active cancer
* Acute infectious disease or history of chronic infections
* Recent (within 3 months) treatment with anabolic steroids, or prolonged systemic corticosteroids.
* Alcohol or drug abuse
* Tobacco use (smoking or chewing)
* Malnutrition (BMI < 18.5 kg/sq meter)
* Obesity (BMI > 30 kg/sq meter)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Change in muscle protein synthesis in response to amino acids | Change from baseline to 3 months
  Measurement of the change in muscle protein synthesis in response to amino acids by standard stable isotope method

SECONDARY OUTCOMES:
Muscle mass | Change from baseline to 3 months
  Measurement in the change in muscle mass by DEXA scan
Muscle function | Change from baseline to 3 months
  Measurement of the change in muscle function by standard methods

CONTACTS AND LOCATIONS:
Overall Officials: Blake B Rasmussen, PhD, Principal Investigator — University of Texas
Locations (1):
- UTMB, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moro T, Brightwell CR, Deer RR, Graber TG, Galvan E, Fry CS, Volpi E, Rasmussen BB. Muscle Protein Anabolic Resistance to Essential Amino Acids Does Not Occur in Healthy Older Adults Before or After Resistance Exercise Training. J Nutr. 2018 Jun 1;148(6):900-909. doi: 10.1093/jn/nxy064. PMID 29796648